CLINICAL TRIAL: NCT06019468
Title: Clinical Study of Envolizumab Combined With Radiotherapy for Neoadjuvant Treatment of Locally Advanced Thymic Cancer
Brief Title: Neoadjuvant Treatment For Locally Advanced Thymic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Deping Zhao, Administrative Director of Thoracic Surgery Department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR005
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Thymic Carcinoma
MeSH Terms: conditions — Thymoma | interventions — Radiotherapy; envafolimab

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant immunotherapy combined with radiotherapy (Experimental): Treatment arms comprise 10-20 cycles of radiotherapy and 2-4 cycles of maintenance therapy with Envolizumab
  Interventions: Other: Envolizumab combined with radiotherapy

INTERVENTIONS:
Other: Envolizumab combined with radiotherapy — Application of Envolizumab combined with radiotherapy for neoadjuvant treatment of locally advanced thymic cancer. Firstly, 20-40Gy radiation therapy was administered 10-20 times. Within one week after the start of radiation therapy, Envolizumab (300 mg, D1, Q3W, subcutaneous injection) was administered. Immunotherapy was maintained for 2-4 cycles, and surgery was performed after evaluation by the attending physician.
  Other Names: KN035

SUMMARY:
The aims of this study are to verify the feasibility, effectiveness, and safety of the combination of enrolizumab and radiotherapy for neoadjuvant treatment for locally advanced thymic carcinoma, and to provide recommendations for the establishment of unified evaluation criteria for the neoadjuvant therapy of thymic cancer by evaluating the pathological remission status of thymic cancer specimens after neoadjuvant treatment.

DETAILED DESCRIPTION:
For patients with locally advanced thymic carcinoma, it is often difficult to perform radical resection. Numerous studies have reported that neoadjuvant therapy can improve the surgical resection rate of thymic tumors by reducing the extent of tumor invasion and eliminating small metastatic lesions, thereby improving patient survival. However, the efficacy of neoadjuvant immunotherapy combined with chemotherapy is limited. This study intends to conduct a single-arm, phase II clinical trial of neoadjuvant immunotherapy combined with radiotherapy for locally advanced thymic carcinoma to verify the feasibility and safety of neoadjuvant immunotherapy combined with radiotherapy. Meanwhile, the investigators evaluate the pathological remission of postoperative specimens to provide recommendations for establishing pathological evaluation criteria for neoadjuvant therapy for thymic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed as thymic carcinoma;
2. Clinical staging III-IVA (TNM staging system), non-myasthenia gravis (MG) patients, expected to undergo surgical resection;
3. On the day when the subject signs the informed consent form, they are ≥ 18 years old and<75 years old, regardless of gender;
4. The subjects are able to understand the informed consent form, voluntarily participate, and sign the informed consent form;
5. Subjects who have not received any anti-thymic tumor treatment in the past, including but not limited to systemic chemotherapy, radiotherapy, or immunotherapy (only those who have received traditional Chinese medicine treatment for anti-tumor indications are allowed to be included, and a cleaning period of at least 2 weeks is required);
6. At least 1 measurable lesion (according to the solid tumor efficacy evaluation standard RECIST V1.1);
7. Physical fitness score of 0 or 1 (ECOG scoring system of the Eastern Cancer Collaborative Group in the United States);
8. Female subjects with fertility must have a negative serum pregnancy test within 7 days before the first administration;
9. Female subjects with fertility or male subjects with partners with fertility agree to use efficient contraceptive measures (with an annual failure rate of less than 1%) from 7 days before the first administration until 24 weeks after the end of administration;
10. The main organ functions within 7 days before the first administration meet the following standards:

    1. Bone marrow function: hemoglobin ≥ 10.0 g/dL (no blood transfusion received within 28 days before hemoglobin test), absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L (no platelet transfusion or IL-11 treatment received within 14 days prior to platelet count test);
    2. Coagulation function: INR and PT<1.5 × ULN, APTT ≤ 1.5 × ULN;
    3. Liver function: transaminases (ALT and AST) ≤ 2.5 × ULN; Total bilirubin ≤ 1.5 × ULN (total bilirubin ≤ 2.5 in subjects with Gilbert's syndrome or liver metastasis) × ULN);
    4. Renal function: serum creatinine clearance rate ≥ 60 mL/min (calculated according to Cockcroft Fault formula);
    5. Adequate lung function: According to the doctor's judgment, lung function can meet the requirements of thymectomy surgery.

Exclusion Criteria:

1. Pathologically confirmed as a thymic neuroendocrine tumor;
2. Subjects who have undergone major surgical treatment (such as abdominal or thoracic surgery; excluding diagnostic puncture or peripheral vascular pathway replacement surgery) or have not recovered from surgical treatment within 28 days before the administration of this trial;
3. Within 14 days before the first administration of this study, systemic corticosteroids (≥ 10 mg/day prednisone, or equivalent amounts of other corticosteroids) or immunosuppressive therapy are required for 7 consecutive days; Excluding inhalation or local application of hormones, or receiving physiological replacement doses of hormone therapy due to adrenal insufficiency; Allow short-term (<7 days) use of corticosteroids for prevention (such as contrast agent allergies) or treatment of non-autoimmune diseases (such as delayed hypersensitivity reactions caused by exposure to allergens);
4. Received live vaccines (including attenuated live vaccines) within 28 days prior to administration in this study;
5. Previously or currently suffering from interstitial pneumonia/lung disease that requires systemic hormone therapy;
6. Previously or currently suffering from autoimmune diseases, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener syndrome (granulomatosis of vasculitis, Graves disease, rheumatoid arthritis, pituitary inflammation, uveitis), autoimmune hepatitis, systemic sclerosis (scleroderma, etc.), Hashimoto's thyroiditis (exceptions see below), autoimmune vasculitis Autoimmune neuropathy (Guillain Barre syndrome), etc. The following cases are excluded: type I diabetes, hypothyroidism with stable hormone replacement therapy (including hypothyroidism caused by autoimmune thyroid disease), psoriasis or vitiligo without systemic treatment;
7. Other malignant tumors were combined within 5 years before the first administration, excluding cured skin squamous cell carcinoma, basal cell carcinoma, non-muscle invasive bladder cancer, localized low-risk prostate (defined as stage ≤ T2a, Gleason score ≤ 6, and PSA ≤ 10ng/mL at the time of diagnosis of prostate cancer (if measured, patients who have received radical treatment and have no PSA biochemical relapse can participate in this study), and in situ cervical/breast cancer;
8. Have uncontrolled heart, kidney, gastrointestinal tract, infectious diseases and other complications;
9. Previous history of allogeneic bone marrow or organ transplantation;;
10. Previously treated with any antibody/drug (immune checkpoint) targeting T cell co-regulatory proteins, such as anti PD (L) 1, CTLA-4, 4-1BB, LAG 3, TIM 3, or anti CD127; Previously received anti-tumor vaccine treatment
11. Previous history of allergic reactions to antibody-based drugs and intolerance (≥ Level 3 NCI-CTCAE V5.0); Any past history of rapid allergic reactions and uncontrollable asthma (i.e. uncontrollable asthma symptoms of 3 or more of the 3 or more characteristics of partially controlled asthma); Previous obvious allergies to drugs (such as severe allergic reactions, immune-mediated hepatotoxicity, immune-mediated thrombocytopenia or anemia);
12. Pregnant and/or lactating women;
13. Other situations that may affect the safety or compliance of drug treatment in this study, including but not limited to mental illness, uncontrolled large amounts of serous fluid accumulation, or subjects who require repeated drainage (recurrence within 2 weeks after intervention) with moderate to large amounts of serous fluid accumulation, cachexia, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate（ORR） | 24 hour
  ORR was defined as the best overall response (BoR), the proportion of participants in complete and partial response among the number of participants in each treatment group who received at least one medication.

SECONDARY OUTCOMES:
Disease control rate（DCR） | 24 hours
  DCR is defined as the proportion of imaging findings of CR, PR, and stable disease (SD) in all subjects evaluated according to RECIST V1.1 after completing neoadjuvant immunotherapy combined with radiotherapy
Radical resection rate（R0） | 24 hours
  Pathological evaluation of the tumor margin, and based on whether the margin is gross or microscopic positive, it is divided into radical resection (R0), microscopic residual lesion (R1), or gross residual lesion (R2)
Pathological remission rate | 7 days
  Conduct pathological evaluation based on postoperative specimens to evaluate the percentage of surviving tumor cells, necrosis, and interstitial components in the original tumor bed area.
disease-free survival（DFS） | 5 years
  The time interval between receiving surgical treatment and tumor recurrence or death due to tumor progression
overall survival（OS） | 5 years
  The time interval between receiving surgical treatment and the patient's death due to any reason, and the patient is still alive during the final follow-up, with the survival time ending at the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Deping Zhao, MD,PhD, Principal Investigator — Shanghai Pulmonary Hospital, School of Medicine, Tongji University
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No